CLINICAL TRIAL: NCT05067023
Title: Evaluation for Benign and Malignant Pulmonary Ground-glass Nodules Based on MRI Dynamic Contrast Enhanced Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, investigator, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QianfoshanH Z
Record Dates: First submitted 2021-09-09; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Nodules
MeSH Terms: conditions — Multiple Pulmonary Nodules | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI scan (Experimental): All participants will undergo 1 DCE-MRI scan before surgery or puncture.
  Interventions: Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: MRI scan — All participants will undergo 1 DCE-MRI scan.

SUMMARY:
Computed tomography (CT) is critical for the diagnosis of lung nodules as well as for therapeutic management. Repeated CT examinations will raise the issue of the cumulative radiation dose and subsequent risk of cancer, thus pushing the need for imaging techniques using low or no radiation dose. Magnetic Resonance Imagery (MRI) with ultrashort echo time (UTE) pulse sequences with high signal-to-noise and spatial resolution is a promising alternative for lung nodules imaging.The purpose of the study is to evaluate the value of dynamic contrast-enhanced MR imaging (DCE-MRI) to discriminate of malignant from benign lesions.

DETAILED DESCRIPTION:
Computed tomography (CT) is critical for the diagnosis of lung nodules as well as for therapeutic management. Repeated CT examinations will raise the issue of the cumulative radiation dose and subsequent risk of cancer, thus pushing the need for imaging techniques using low or no radiation dose. Magnetic Resonance Imagery (MRI) with ultrashort echo time (UTE) pulse sequences with high signal-to-noise and spatial resolution is a promising alternative for lung nodules imaging.The purpose of the study is to evaluate the value of DCE-MRI to discriminate of malignant from benign lesions.In this study, the investigators are going to validate the efficacy of the DCE-MRI for diagnosing early lung cancer by comparing results of the pre-surgery MRI imaging with the post-surgery pathology.

ELIGIBILITY:
Inclusion Criteria:

* Ground-glass pulmonary nodules found by CT scan
* Plan to accept surgery or puncture due to the pulmonary nodules
* Absence of treatment such as chemotherapy or radiotherapy and biopsy
* Adequate renal function to tolerate intravenous gadolinium
* Agree to sign informed consent
* Able to lie still during DCE-MRI

Exclusion Criteria:

* Fail to understand or agree to sign informed consent
* Implanted pacemaker or cardiac defibrillator
* Contraindications to undergoing MRI
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-20 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Volume transfer constant (Ktrans) | 12 months
  Pharmacokinetic parameters will be estimated by fitting a pharmacokinetic model to the actual time-intensity curves obtained from the DCE-MRI.
the fractional volume of extravascular extracellular space of the target tissue (ve) | 12 months
  Pharmacokinetic parameters will be estimated by fitting a pharmacokinetic model to the actual time-intensity curves obtained from the DCE-MRI.
the rate constant (kep) | 12 months
  Pharmacokinetic parameters will be estimated by fitting a pharmacokinetic model to the actual time-intensity curves obtained from the DCE-MRI.